CLINICAL TRIAL: NCT05442723
Title: Extensively Diseased Left Anterior Descending Coronary Artery: On Pump vs Off Pump CABG?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kareem Ahmed Hosny, Principle investigator, Assiut University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AssiutMed
Record Dates: First submitted 2022-02-26; First posted 2022-07-05 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: CAD - Coronary Artery Disease
Keywords: On-pump; off-pump; CABG; LAD
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case (Other): Patients with extensive LAD disease treated with off-pump CABG
  Interventions: Procedure: Off-Pump CABG
- Control (Other): Patients with extensive LAD disease treated with on-pump CABG
  Interventions: Procedure: On-Pump CABG

INTERVENTIONS:
Procedure: On-Pump CABG — coronary artery grafting by using cardiopulmonary bypass machine
  Other Names: CABG
  Arms: Control
Procedure: Off-Pump CABG — coronary artery grafting by beating heart technique
  Arms: Case

SUMMARY:
Diseased left Anterior descending coronary artery (LAD) is one of the most challenging conditions in Bypass surgery. we investigate whether on-pump coronary artery bypass grafting (CABG) is more beneficial in those critical patients or off-pump surgery.

ELIGIBILITY:
Inclusion Criteria:

* any patient with diffuse LAD disease indicated for open heart surgery

Exclusion Criteria:

* no concomitant valve disease
* any patient can be treated by medical treatment or PCI

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-02-25 (Actual); Primary Completion 2023-02-24 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
mortality | 30 days post operative
  follow up post-operative track of the patient for any noticed mortality rate
Morbidity | 60 days post operative
  follow up post-operative track of the patient for any noticed complications

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university heart hospital, Asyut, Egypt